CLINICAL TRIAL: NCT02824484
Title: Promoting Post-traumatic Growth in Cancer Patients: a Study Protocol for a Randomized Controlled Trial of Guided Written Disclosure
Brief Title: A Guided Written Disclosure Intervention to Promote Post-traumatic Growth in Cancer Patients GUIDED WRITTEN DISCLOSURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: European University of Rome (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2015/0024360
Record Dates: First submitted 2016-06-10; First posted 2016-07-06 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: Guided written disclosure protocol; Emotional disclosure; Meaning; Post-Traumatic Growth; Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided Written Disclosure Protocol (Experimental): GWDP consists of three 20-minutes writing sessions. Participants write every two weeks at home following the specific instructions for each session.
  Interventions: Behavioral: GWDP
- Control (Placebo Comparator): Control condition consists of three 20-minutes writing sessions. Participants write every two weeks at home following the instructions. Their task is constructed to be emotionally neutral.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: GWDP — In each writing session participants are asked to:
  1. Describe memories concerning cancer illness in a chronological order, with an objective and detached attitude
  2. Describe: (a) thoughts and emotions perceived during the illness experience; (b) the impact of illness on their daily lives, and how it has changed their attitudes toward life.
  3. Focus on their actual situation, think about the entire illness experience, and report on the following aspects: -Their present thoughts and feelings, and how those differ from the ones felt during the illness experience. -To what extent they have come to terms with, understand and appreciate themselves to have dealt successfully with the illness.
  Other Names: Guided Written Disclosure Protocol
  Arms: Guided Written Disclosure Protocol
Behavioral: Control — Participants are requested to write about events of their daily routine happened during the past week; they are also asked to focus on facts, with an objective and detached attitude.
  Arms: Control

SUMMARY:
This study aims to investigate the efficacy of Guided Written Disclosure Protocol (GWDP) in promoting post-traumatic growth through a process of meaning reconstruction in cancer patients at the end of chemotherapy. Also, the intervention (GWDP) intends to reduce distress symptoms (i.e. intrusive thoughts, avoidance, depression and anxiety).

DETAILED DESCRIPTION:
Study aims The primary aim of this study is to assess the efficacy of the Guided Written Disclosure Protocol in promoting post-traumatic growth in stage I-III breast and colon cancer patients at the end of their adjuvant chemotherapy.

The secondary aims of the study include

* Evaluating the efficacy of the GWDP in terms of intrusive thoughts and avoidance reduction
* Assessing the efficacy of the GWDP in terms of reduction of depression and anxiety
* Investigating the relationship between constructed meaning and post-traumatic growth.

Methods Study design The study is a randomized controlled trial. Eligible patients who give their consent to participate in the study will be randomized to receive the GWDP intervention (experimental group) or a control intervention (control group).

Participants Participants will be recruited in the Oncological Day Hospitals (DH) of the Scientific Research and Care Institute (IRCCS) Santa Maria Nuova Hospital of Reggio Emilia - Oncology Unit

Eligibility criteria will be assessed by reviewing the patients' medical record and verified at the time of recruitment.

Randomization Eligible patients, who agree to participate in the study, will be randomly assigned to the GWDP condition or to the control condition with an allocation ratio 1:1, stratified by the oncological DH. Randomization is carried out through a central phone randomization center using computer generated random numbers.

After the registration of the patient basic information, the trial center will attribute a unique code to the included patient, and communicate to the professional the allocated condition. This code will be reported in all the forms related to each patient.

The interventions The experimental intervention (GWDP) consists of three 20-minutes writing sessions in which instructions are provided to patients that have experienced the traumatic event of cancer diagnosis and therapies. Initially, participants are invited to recall chronologically the facts concerning the traumatic event, and then to label the emotions related to those facts, appraise immediate changes in priorities, reflect on their current feelings, and on coping mechanisms they have learned. Moreover, they are asked to reflect on how the experience of cancer has changed their view about life and themselves, teaching them to cope with other difficulties that may arise in the future.

Below, investigators report a synthesis of the tasks concerning each of the three writing sessions. Participants are asked to:

1. describe memories concerning cancer illness in a chronological order, with an objective and detached attitude.
2. describe: (a) thoughts and emotions perceived during the illness experience; (b) the impact of illness on their daily lives, and how it has changed their attitudes toward life.
3. focus on their actual situation, think about the entire illness experience, and report on the following aspects:

   * their present thoughts and feelings, and how those differ from the ones felt during the illness experience.
   * to what extent they have come to terms with, understand and appreciate themselves to have dealt successfully with the illness.
   * what they have learned from illness in terms of personal insights, knowledge and skills, and how these resources could be useful in their future.
   * how they will cope with other similar events in the future.

Participants are asked to find a quiet place and time in their home to write without being disturbed. The first writing session will be performed by two weeks from the initial assessment (T0), and the following two sessions once every two weeks.

Original instructions were translated into Italian, and adapted to the specific traumatic experience of cancer diagnosis and treatment.

The control condition consists of three 20-minutes writing sessions in which participants are requested to write about events of their daily routine happened during the past week; they are also asked to focus on facts, with an objective and detached attitude. An active control intervention is used to account for both general (i.e., due to a written general description) and specific effects (i.e., due to a written emotional expression, together with a cognitive reframing) of the writing task.

As for the experimental group, participants are asked to find a quiet place and time to write without being disturbed. It was used the same time interval between sessions as for the GWDP.

One day before each writing session, patients in both conditions will be contacted on the telephone by the researcher, who will check their understanding of instructions included in the booklet, and remind them to perform the writing task. Failure to contact the patient will be recorded in the patient form.

Procedures of recruitment and assessment Recruitment and baseline assessment (T0). One or more health care professionals (oncologists, nurses or psychologists) will participate as recruiters and evaluators. They will be trained by the Steering Committee about study aims and procedures, and provided with study materials. The preferred method of recruitment involves the oncologist in informing eligible patients, who attend DH for their medical consultation. In case of impediments to recruitment (e.g., oncologists' lack of motivation for involvement in the study, medical consultation scheduled beyond eight months after the end of chemotherapy, patients' unavailability at the time of medical appointment), a letter will be sent to eligible patients presenting general information about the study. Three to seven days later, a member of the study staff will call the patient by phone to give further information, and to verify his/her availability to participate.

Patients interested in the intervention will meet a health care professional, who will explain both the study aims and the writing tasks, providing them with the information sheet, and collecting socio-demographic data and health information (i.e., age, sex, educational level, marital status, time since diagnosis, disease site and stage, and treatment received). Patients, who agree to participate, will give their written consent. The health care professional will administrate baseline questionnaires, and then will contact the trial center for randomization. Finally, the booklet concerning the intervention, according to allocation group, will be provided to the participant. Anonymity will be guaranteed for both written texts and outcomes assessment.

Post-intervention and follow- up assessments (T1 and T2). Participants will be re-assessed for the study outcomes three months after baseline (T1), with a time tolerance of ± 15 days, whenever is possible during any medical consultation. In this occasion, the booklet containing the patient's written texts will be returned. Follow-up evaluation (T2) will be performed six months after the post-intervention assessment (with the same time tolerance of ± 15 days), whenever is possible during any medical consultation.

Hypotheses Main hypothesis. Investigators expect that, after the intervention, participants in the GWDP group will have higher scores on the Post-Traumatic Growth Inventory as compared to the control group.

Meaning construction is deemed as the mechanism underlying the restructuring of more adaptive schemas that lead to growth. Therefore, investigators expect that increased levels of PTG could be moderated by constructed meaning, measured by the Constructed Meaning Scale.

Secondary hypothesis. Investigators hypothesize that, after the intervention, participants in the GWDP group will have lower scores on the Impact of Events Scale as compared to the control group. Investigators also predict that participants in the GWDP group will have lower scores on the Hospital Anxiety and Depression Scale as compared with the control group.

Sample size A prospective power analysis revealed that the current study would require 250 participants to achieve 80% power. The predicted effect size (Hedges's g = 0.36) is estimated according to a recent meta-analysis on the effect of psychological interventions on post-traumatic growth.

Data analysis A preliminary analysis will be performed to compare, at baseline, the differences of clinical and demographic data between the two groups (GDWP intervention vs. control intervention). After that, a 2 X 3 mixed factorial design ANOVA will be performed for each dependent variable (Post-traumatic growth, and distress measures). The "between" factor is intervention with two levels (yes/no) and the "within" factor is time with three levels (T0/T1/T2). Adjusted analysis of variance with sociodemographic and health variables as covariant will be performed. Finally, the potential moderating role of constructed meaning on the effect of GWDP will be according to the MacArthur approach.

Ethical issues The data collection and the intervention will be performed in accordance with the ethical standards of the local Ethical committee, which have approved the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. A histologically-confirmed stage I-III breast or colon cancer
2. Adjuvant chemotherapy completed by no more than eight months
3. Disease free (no evidence of metastatic disease) according to what reported by the oncologist during the follow-up oncological consultation
4. Aged 18 years or over
5. Property of written and spoken Italian language

Exclusion Criteria:

1. Having received a structured psychological intervention performed by a psychologist or by a psychiatrist, for at least six months during the last three years
2. Having received a psychopharmacological treatment for a codified psychiatric disorder (according to the DSM-V) during the last three years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in post-traumatic growth from baseline to post-intervention assessment and at 6 months follow-up. Post-Traumatic Growth Inventory (PTGI) will be used to assess this outcome | Baseline (T0): before randomization. Post-intervention (T1): three months (plus or minus 15 days) from (T1). Follow-up (T2): six months after T1.
  21-item questionnaire

SECONDARY OUTCOMES:
Change in constructed meaning from baseline to post-intervention assessment and at 6 monts follow-up. Constructed Meaning Scale (CMS) will be used to assess this outcome | Baseline (T0): before randomization. Post-intervention (T1): three months (plus or minus 15 days) from (T1). Follow-up (T2): six months after T1.
  8-item questionnaire
Change in intrusive thoughts and avoidance from baseline to post-intervention assessment and at 6 months follow-up. Impact of Event Scale (IES) will be used to assess this outcome | Baseline (T0): before randomization. Post-intervention (T1): three months (plus or minus 15 days) from (T1). Follow-up (T2): six months after T1.
  15-item questionnaire
Change in anxiety and depression from baseline to post-intervention assessment and at 6 months follow-up. Hospital Anxiety and Depression Scale (HADS) will be used to assess this outcome | Baseline (T0): before randomization. Post-intervention (T1): three months (plus or minus 15 days) from (T1). Follow-up (T2): six months after T1.
  14.item questionnaire

OTHER OUTCOMES:
Expectancy about change in personal growth as a result of the intervention (Treatment Expectancy, TE) | baseline (T0)
  1 item asking patients to what extent they expect improvement in personal growth after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Arcispedale S. Maria Nuova-IRCCS, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: Undecided